CLINICAL TRIAL: NCT05106842
Title: Hydrotherapy Versus Classical Rehabilitation After Surgical Rotator Cuff Repair: a Randomized Prospective Study
Brief Title: Hydrotherapy Versus Classical Rehabilitation After Surgical Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Sponsor-Investigator, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LaTourH
Record Dates: First submitted 2021-08-18; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: This prospective case-control clinical study is randomized 1:1 between rehabilitation with hydrotherapy and land-based rehabilitation.
Who Masked: Outcomes Assessor
Masking Description: Medical history, demographics, and clinical scores will be collected by the selected and blinded investigator (on corresponding case reporting forms). Patients will be informed of the blinding procedure. They should not unblind investigator during the whole follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrotherapy after Rotator Cuff Repair (Active Comparator): The participants will start with passive mobilization right after surgery for 4 weeks. Intervention in hydrotherapy will follow after that.
  Interventions: Other: Hydrotherapy
- Classical Land Based Rehabilitation after Rotator Cuff Repair (Active Comparator): The participants will start with passive mobilization right after surgery for 4 weeks. Intervention in classic dry land based rehabilitation will follow after that.
  Interventions: Other: Land-based Therapy

INTERVENTIONS:
Other: Hydrotherapy — Aquatic therapy was performed in a swimming pool (depth 125-140 cm, temperature 28-31°C) supervised by a physiotherapist. Patients were asked to kneel or sit to submerge both shoulders to perform exercises consisting of progressive passive and active motion of the shoulder for 4-6 weeks, then strengthening exercises in a swimming pool for 2-4 months.
  Arms: Hydrotherapy after Rotator Cuff Repair
Other: Land-based Therapy — Land-based therapy was performed at a rehabilitation center supervised by a physiotherapist. Patients performed progressive passive and active-assisted motion of the shoulder for 4-6 weeks, then strengthening exercises for 2-4 months.
  Arms: Classical Land Based Rehabilitation after Rotator Cuff Repair

SUMMARY:
Postoperative rehabilitation following rotator cuff repair is important to promote tendon healing, restore strength, and recover normal function. The aim of this study is to assess whether aquatic rehabilitation is more efficient than classical rehabilitation (land-based session) in term of range of motion, function, and pain than classical rehabilitation (land-based session) after an arthroscopic repair of the rotator cuff.

DETAILED DESCRIPTION:
Introduction:

Postoperative rehabilitation following rotator cuff repair is important to promote tendon healing, restore strength, and recover normal function. Aquatic rehabilitation in hot water allows body relaxation and well-being that promote patient conditioning for efficient rehabilitation and is appreciated by patients. The aim of this study is to assess whether aquatic rehabilitation is more efficient than classical rehabilitation (land-based session) in term of range of motion, function, and pain after an arthroscopic repair of the rotator cuff.

Methods:

This prospective case-control clinical study is randomized 1:1 between rehabilitation with hydrotherapy and land-based (standard) rehabilitation. This superiority trial that included 84 patients that have benefited from an arthroscopic superior cuff repair. Patients were evaluated clinically at 6 weeks, 3, 6 and 24 months and using ultrasound at 6 months. Multivariable linear regressions were performed to determine if 2-year postoperative scores were associated with gender, body mass index (BMI), age at index operation, rehabilitation group (Hydrotherapy vs Standard), and baseline passive range of motion (PROM) Active range of motion (AROM).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Arthroscopic cuff repair of supraspinatus tendon (with potentially concomitant of infraspinatus tendon repair, tenodesis or tenotomy of brachial biceps tendon, acromioplasty, and distal clavicle removal).

Exclusion Criteria:

* Lesion of subscapularis tendon;
* SLAP lesion;
* Second rotator cuff surgery;
* Frozen shoulder (i.e. Forward flexion reduced of 25% or more);
* Inability to follow the study protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Passive forward flexion | 1.5 months
  As primary outcome, we will evaluate if passive antepulsion is superior with balneotherapy than classical rehabilitation (land-based session). We consider the effective intervention with a 105 ° forward flexion.

SECONDARY OUTCOMES:
Pain (Visual Analogue Scale) | 1.5 months
  Minimum score is 0 while maximum score is 10. The higher the score, the worse is the outcome.
Constant Score | 1.5 months
  Minimum score is 0 while maximum score is 100. The higher the score, the better is the outcome.
Single Assessment Numeric Evaluation (SANE) score | 1.5 months
  Minimum score is 0 while the maximum score is 100. The higher the score, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brady B, Redfern J, MacDougal G, Williams J. The addition of aquatic therapy to rehabilitation following surgical rotator cuff repair: a feasibility study. Physiother Res Int. 2008 Sep;13(3):153-61. doi: 10.1002/pri.403. PMID 18548557
- [Background] Burmaster C, Eckenrode BJ, Stiebel M. Early Incorporation of an Evidence-Based Aquatic-Assisted Approach to Arthroscopic Rotator Cuff Repair Rehabilitation: Prospective Case Study. Phys Ther. 2016 Jan;96(1):53-61. doi: 10.2522/ptj.20140178. Epub 2015 Jul 23. PMID 26206216
- [Background] Chae CS, Jun JH, Im S, Jang Y, Park GY. Effectiveness of Hydrotherapy on Balance and Paretic Knee Strength in Patients With Stroke: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2020 May;99(5):409-419. doi: 10.1097/PHM.0000000000001357. PMID 31764223
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Cuesta-Vargas AI, Cano-Herrera C, Formosa D, Burkett B. Electromyographic responses during time get up and go test in water (wTUG). Springerplus. 2013 May 10;2(1):217. doi: 10.1186/2193-1801-2-217. Print 2013 Dec. PMID 23705108
- [Background] Ghodadra NS, Provencher MT, Verma NN, Wilk KE, Romeo AA. Open, mini-open, and all-arthroscopic rotator cuff repair surgery: indications and implications for rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):81-9. doi: 10.2519/jospt.2009.2918. PMID 19194025
- [Background] Giaquinto S, Ciotola E, Dall'Armi V, Margutti F. Hydrotherapy after total knee arthroplasty. A follow-up study. Arch Gerontol Geriatr. 2010 Jul-Aug;51(1):59-63. doi: 10.1016/j.archger.2009.07.007. Epub 2009 Sep 6. PMID 19735951
- [Background] Gilbart MK, Gerber C. Comparison of the subjective shoulder value and the Constant score. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):717-21. doi: 10.1016/j.jse.2007.02.123. PMID 18061114
- [Background] Kukkonen J, Kauko T, Vahlberg T, Joukainen A, Aarimaa V. Investigating minimal clinically important difference for Constant score in patients undergoing rotator cuff surgery. J Shoulder Elbow Surg. 2013 Dec;22(12):1650-5. doi: 10.1016/j.jse.2013.05.002. Epub 2013 Jul 12. PMID 23850308
- [Background] Longo UG, Berton A, Risi Ambrogioni L, Lo Presti D, Carnevale A, Candela V, Stelitano G, Schena E, Nazarian A, Denaro V. Cost-Effectiveness of Supervised versus Unsupervised Rehabilitation for Rotator-Cuff Repair: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2020 Apr 21;17(8):2852. doi: 10.3390/ijerph17082852. PMID 32326198
- [Background] Mazzocca AD, Arciero RA, Shea KP, Apostolakos JM, Solovyova O, Gomlinski G, Wojcik KE, Tafuto V, Stock H, Cote MP. The Effect of Early Range of Motion on Quality of Life, Clinical Outcome, and Repair Integrity After Arthroscopic Rotator Cuff Repair. Arthroscopy. 2017 Jun;33(6):1138-1148. doi: 10.1016/j.arthro.2016.10.017. Epub 2017 Jan 19. PMID 28111006
- [Background] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Background] Patte D. Classification of rotator cuff lesions. Clin Orthop Relat Res. 1990 May;(254):81-6. PMID 2323151
- [Background] Rahmann AE, Brauer SG, Nitz JC. A specific inpatient aquatic physiotherapy program improves strength after total hip or knee replacement surgery: a randomized controlled trial. Arch Phys Med Rehabil. 2009 May;90(5):745-55. doi: 10.1016/j.apmr.2008.12.011. PMID 19406293
- [Background] Speer KP, Cavanaugh JT, Warren RF, Day L, Wickiewicz TL. A role for hydrotherapy in shoulder rehabilitation. Am J Sports Med. 1993 Nov-Dec;21(6):850-3. doi: 10.1177/036354659302100616. No abstract available. PMID 8291638
- [Background] Thomson S, Jukes C, Lewis J. Rehabilitation following surgical repair of the rotator cuff: a systematic review. Physiotherapy. 2016 Mar;102(1):20-8. doi: 10.1016/j.physio.2015.08.003. Epub 2015 Sep 8. PMID 26510584
- [Background] Williams GR Jr, Rockwood CA Jr, Bigliani LU, Iannotti JP, Stanwood W. Rotator cuff tears: why do we repair them? J Bone Joint Surg Am. 2004 Dec;86(12):2764-76. No abstract available. PMID 15590865